CLINICAL TRIAL: NCT00507715
Title: Clinical Trial to Study the Modification of the Pharmacokinetic Profile of Levodopa by the Fiber Plantago Ovata Husk
Brief Title: Study of the Modification of the Pharmacokinetic Profile of Levodopa by the Fiber Plantago Ovata Husk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PLAN-EC-LDOPA-FI; EudraCT number:2006-000491-33
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: Parkinson's Disease, Idiopathic
Keywords: Parkinson's Disease, Idiopathic; l-dopa levels; plantago ovata husk
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Plantago ovata husk
  Interventions: Drug: Plantago ovata husk
- 2 (Placebo Comparator): hemicellulose crystalline
  Interventions: Other: hemicellulose crystalline

INTERVENTIONS:
Drug: Plantago ovata husk — 5 g of effervescent powder (3.5 g pf plantago ovata husk) t.i.d. during 14 days
  Arms: 1
Other: hemicellulose crystalline — 5g effervescent powder t.id. during 14 days
  Arms: 2

SUMMARY:
The purpose of this trial is to study the effect of the association levodopa/carbidopa with plantago ovata husk in Parkinson´s disease patients of recent diagnostic, that are being treated with levodopa/carbidopa.

DETAILED DESCRIPTION:
Although the treatment with l-dopa is the election treatment for Parkinson´s disease, a high number of patients develop motor complications, including, fluctuations and dyscinesia after some years of treatment.

The origin of the fluctuations is not well established, but it could be attributed, al least partially, a pharmacokinetics factors. So that, it could improve the answer and reduce the adverse reaction if we reach more stable levels of L-dopa in the circulation. The first experimental studies in animals showed that Plantago ovata husk has an influence in the pharmacokinetics parameters of L-dopa, obtaining more stable levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnostic of idiopathic Parkinson disease, with well controlled symptomatology with administration of l-dopa/carbidopa.
* At least 3 months of treatment continued of levodopa.
* Patients that give the their consent to participate in the study.

Exclusion Criteria:

* Patients with diagnostic of idiopathic Parkinson disease, with bad controlled symptomatology with administration of l-dopa/carbidopa.
* Patients with allergic predisposition to Plantago ovata husk or other contraindications for its use.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To study how the fiber Plantago ovata husk modifies the pharmacokinetics parameters of the absorption and elimination of L-dopa. | 14 days

SECONDARY OUTCOMES:
To evaluate if the treatment with Plantago ovata husk modifies the biochemical parameters as total cholesterol, HDL y LDL, glycaemia, etc. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sierra Matilde, Ph, phD, Study Chair — Departamento de Ciencias Biomédicas de la Facultad de Veterinaria de la Universidad de León, León (Spain); Carriedo Demetrio, MD, Principal Investigator — Hospital de León, León (Spain)
Locations (1):
- Hospital de León, León, León, Spain